CLINICAL TRIAL: NCT07109739
Title: Dose-Response Effects of Inspiratory Muscle Strength Training on Blood Pressure and Vascular Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00025718
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Systolic Hypertension; Brachial Artery Flow-mediated Dilation
MeSH Terms: conditions — Isolated Systolic Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- 15 Breaths/ Day (Active Comparator): All sessions will be performed at 75% of each participant's PI max 7 days per week, for 6 weeks, using the POWERbreathe K5 device. Each session will take approximately 3-10 minutes depending on the assigned dose group.
  Interventions: Device: POWERbreathe K5
- 30 Breaths/ Day (Active Comparator): All sessions will be performed at 75% of each participant's PI max 7 days per week, for 6 weeks, using the POWERbreathe K5 device. Each session will take approximately 3-10 minutes depending on the assigned dose group.
  Interventions: Device: POWERbreathe K5
- 45 Breaths/ Day (Active Comparator): All sessions will be performed at 75% of each participant's PI max 7 days per week, for 6 weeks, using the POWERbreathe K5 device. Each session will take approximately 3-10 minutes depending on the assigned dose group.
  Interventions: Device: POWERbreathe K5

INTERVENTIONS:
Device: POWERbreathe K5 — The POWERbreathe K5 is portable, battery-powered, and commercially available. No modifications to the FDA-approved design are being made. Its use in this study is consistent with prior published human research and does not constitute a significant deviation from labeled use in terms of safety or function.

SUMMARY:
This study will assess the dose-response effects of Inspiratory Muscle Strength Training (IMST) in adults with above-normal systolic blood pressure over a 6-week period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Resting SBP ≥120 mmHg as measured during screening 1 & 2
* Free from serious CV or metabolic diseases as identified by self-report and blood chemistry analysis.
* No contraindications to IMST (recent abdominal surgery, ruptured eardrum, asthma with very low symptom perception, fractured ribs, or pneumothorax)
* Language: English-speaking, with ability to comprehend study materials and instructions.
* Pre-visit Compliance: Willing to comply with pre-visit instructions (avoiding food and caffeine ≥ 3 hours, vigorous exercise, alcohol, and non-prescribed medications ≥ 24 hours) prior to each measurement visit.
* Lifestyle: Non-smokers (defined as self-report of not smoking cigarettes or vaping over the past year).

Exclusion Criteria:

* Self-report of history of cardiovascular disease, or conditions affecting the ear (e.g., ruptured eardrum).
* Recent abdominal surgery or presence of an abdominal hernia.
* Asthma with very low symptom perception, frequent severe exacerbations, or abnormally low perception of dyspnea.
* Ruptured eardrum or any other condition of the ear.
* Markedly elevated left ventricular end-diastolic volume and pressure.
* Current respiratory conditions such as a cold, sinusitis, or respiratory tract infection (participants may be included once they recover from the respiratory condition).
* Female-Specific: Pregnant or planning to become pregnant during the study period.
* Compliance: Unable or unwilling to comply with pre-visit restrictions (e.g., avoiding caffeine, alcohol, and exercise within specified hours before visits).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure at 6 Weeks | Week 6
  To determine resting SBP before and after 6 weeks of IMST 15, IMST 30, or IMST 45 (75% PI max for all groups) in men and women aged ≥18 years with resting SBP ≥120 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Craighead, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No